CLINICAL TRIAL: NCT03285828
Title: Optimising the Relationship Between Medical Students and Patients Through a Motivational Interviewing Training Programme: a Pilot Pre-post Study
Brief Title: Motivational Interviewing Training for Medical Students: a Pilot Pre-post Study
Acronym: FEMEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bicetre Hospital (Other)
Collaborators: INSERM SC10-US19 (Unknown); University of Paris 5 - Rene Descartes (Other)
Responsible Party: Principal Investigator, DR ANTOINE CHERET, Doctor ANTOINE CHERET, Bicetre Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FEMEM
Record Dates: First submitted 2017-09-08; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Change; Personality, Due to General Medical Condition
Keywords: medical education, motivational interviewing, medical empathy

STUDY DESIGN:
Intervention Model Description: A pilot pre-post study investigating the effects of a training programme, by comparing performance before and after its implementation
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First group (Other): Students received three four-hour sessions of a basic motivationnal interviewing training over a one week period. The students interviewed for 15 minutes a caregiver playing the role of a patient, six weeks before and three weeks after the training.
  Interventions: Behavioral: motivationnal interviewing training
- Second group (Other): Students received three four-hour sessions of a basic motivationnal interviewing training over a one week period. The students interviewed for 15 minutes a caregiver playing the role of a patient, six weeks before and three weeks after the training.
  Interventions: Behavioral: motivationnal interviewing training

INTERVENTIONS:
Behavioral: motivationnal interviewing training — The students received three four-hour sessions of basic motivationnal interviewing training :
  1. Viewing and commenting on video clips illustrating motivational and non-motivational doctor-patient interactions.
  2. Lectures and the distribution of memory aids.
  3. Practical exercises: making "reflections", asking open questions; exploring ambivalence; dealing with resistance; expressing empathy, summarising.
  4. Role-playing, based on several situations, each involving two students. The investigators deliberately chose a non-medical situation (conflict between a mother and a student asking her for pocket money to go out for fun, the day before a university examination) for the first situation. All the other situations concerned changes to healthier behaviour in a medical setting, but with a goal different from that used for the first or the second simulated interview before motivationnal interviewing training.

SUMMARY:
Objective is to evaluate the impact of a basic training programme in motivational interviewing (MI) for medical students, by comparing the ability of students to promote behavioural changes through relationship skills and to conduct a motivational interview before and after training.

DETAILED DESCRIPTION:
Design: A pilot pre-post study in 20 students by comparing students' performance before and after MI training session.

Setting: Bicêtre Hospital, Assistance Publique Hôpitaux de Paris, France.

Interventions: Students received three four-hour sessions of a basic MI training over a one week period. The students interviewed for 15 minutes a caregiver playing the role of a patient, six weeks before and three weeks after the training.

Main outcome measures: Global scores by two independent raters who used the Motivational Interviewing Treatment Integrity (MITI) 3.1.1 code, perception of student's empathy by the caregivers (CARE questionnaire), self-efficacy of students to engage in a patient-centred relationship (SEPCQ score), and student's satisfaction with the odds of achieving the target goal.

ELIGIBILITY:
Inclusion Criteria:

* Students in clinical internships (fourth or fifth year of medical courses) in the Immunology-Infection-Inflammation-Endocrinology Division of Bicêtre Hospital, Assistance Publique Hôpitaux de Paris.
* signed consent

Exclusion Criteria:

* participation refused
* prior training in motivational interviewing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
GLOBAL MITI scores (MITI = Motivational Interviewing Treatment Integrity version 3.1.1) | 15 mn
  Global scores by two independent raters who used the Motivational Interviewing Treatment Integrity (MITI) 3.1.1 code
perception of student's empathy by the caregivers | 15 mn
  CARE questionnaire (CARE = The Consultation And Relational Empathy questionnaire)
self-efficacy of students to engage in a patient-centred relationship | 15 mn
  SEPCQ score (SEPCQ = The self-efficacy in patient-centeredness score)
student's satisfaction with the odds of achieving the target goal. | 15 mn
  specific questionnary (Analog scale of satisfaction from 1 (not satisfied) to 10 (very statisfied))

CONTACTS AND LOCATIONS:
Overall Officials: ANTOINE CHERET, Principal Investigator — Bicetre Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rollnick S, Butler CC, Kinnersley P, Gregory J, Mash B. Motivational interviewing. BMJ. 2010 Apr 27;340:c1900. doi: 10.1136/bmj.c1900. No abstract available. PMID 20423957